CLINICAL TRIAL: NCT00874094
Title: Pilot Evaluation of Platelet Rich Fibrin Matrix (PRFM) for the Correction of Nasolabial Folds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08.01
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Nasolabial Folds
Keywords: nasolabial folds; platelet rich plasma; fibrin matrix; facial rhytids; dermal filler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- platelet rich fibrin matrix (Active Comparator): Both nasolabial folds treated with 0-2 cc of autologous platelet rich fibrin matrix,sufficient to efface nasolabial fold
  Interventions: Biological: Platelet rich fibrin matrix

INTERVENTIONS:
Biological: Platelet rich fibrin matrix — 0-2 cc of autologous platelet rich fibrin matrix injected intra and subdermally to effect nasolabial fold.

SUMMARY:
Platelets are a component of blood, which contain factors which can enhance wound healing. This study proposes to evaluate the clinical response of laugh lines treated with a concentrated preparation of the subject's own platelets injected into or under the skin by taking serial photographs of the subject's face over a 12 week period. Also, the same preparation will be injected into or under the skin of the arm near the elbows, and serial biopsies will be taken over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* aged 25- 75 years
* with moderate to severe nasolabial folds

Exclusion Criteria:

* pregnant
* allergy to local anesthetics
* history of bleeding disorder
* active infection at the treatment site
* injectable filler in the nasolabial folds within past year

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sclafani, MD, Principal Investigator — The New York Eye & Ear Infirmary
Locations (1):
- The New York Eye & Ear Infirmary- Otolaryngology Faculty practice satellite, Chappaqua, New York, United States

REFERENCES:
- [Result] Sclafani AP. Platelet-rich fibrin matrix for improvement of deep nasolabial folds. J Cosmet Dermatol. 2010 Mar;9(1):66-71. doi: 10.1111/j.1473-2165.2010.00486.x. PMID 20367676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with moderate to severe nasolabial folds were included.
Pre-assignment Details: Any patient who refused to attend all scheduled follow up visits were to be excluded.
Groups:
- Treatment With Platelet Rich Fibrin Matrix: Both nasolabial folds treated with platelet rich fibrin matrix
Period: Overall Study
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 54.27 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Difference in Wrinkle Assessment Score, Between Pre-treatment and 12 Weeks Post-treatment.
Description: Difference in wrinkle assessment score, values ranging from 0 (least noticeable) to 5 ( most noticeable) (scores on a scale)between pre-treatment and 12 weeks post-treatment.
Time Frame: Difference in Measurements taken Pre-treatment and 12 weeks after treatment.
Population: Number of participants were calculated based on need to achieve 1 unit improvement of Wrinkle Assessment score over baseline (pre-treatment) to be clinically relevant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Number analyzed (Participants) | 15
units on a scale | 1.13 (0.76)

2. Secondary Outcome: Difference in Wrinkle Assessment Scores Between Pre-treatment and 1 Week
Description: Difference in Wrinkle Assessment Scores, values ranging from 0 (least noticeable) to 5 ( most noticeable) (scores on a scale), between Pre-treatment and 1 week
Time Frame: pre-treatment to 1 week after treatment
Population: The number of participants required to demonstrate a 1 point difference between pre and post treatment values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Number analyzed (Participants) | 15
units on a scale | .65 (.68)

3. Secondary Outcome: Difference in Wrinkle Assessment Score Between Pretreatment and 2 Weeks
Description: Difference in Wrinkle Assessment Scores, values ranging from 0 (least noticeable) to 5 ( most noticeable) (scores on a scale), between Pre-treatment and 2 weeks
Time Frame: Pre-treatment to 2 weeks after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Number analyzed (Participants) | 15
units on a scale | .97 (.75)

4. Secondary Outcome: Difference in Wrinkle Assessment Score Between Pretreatment and 6 Weeks
Description: Difference in Wrinkle Assessment Scores, values ranging from 0 (least noticeable) to 5 ( most noticeable) (scores on a scale), between Pre-treatment and 6 Weeks
Time Frame: Pre-treatment to 6 weeks after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Number analyzed (Participants) | 15
units on a scale | 1.08 (.59)

ADVERSE EVENTS:
Arm/Group | Treatment With Platelet Rich Fibrin Matrix
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No